# Cover Page for Protocol

| Sponsor name: | Catalyst Pharmaceuticals, Inc. |
|---|---|
| NCT number | 03579966 |
| Sponsor trial ID | MSK-003 |
| Official title of study | Long Term Safety Study of Amifampridine Phosphate in Patients with MuSK Antibody |
| | Positive and AChR Antibody Positive |
| | Myasthenia Gravis Patients |
| Document date | 15 Oct 2021 |

# **Statistical Analysis Plan (SAP)**

Study No. MSK-003

# Long Term Safety Study of Amifampridine Phosphate in Patients with MuSK Antibody Positive and AChR Antibody Positive Myasthenia Gravis Patients

Version 1.0

October 15, 2021

Prepared for Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134

Prepared by STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 www.statkingclinical.com



# **Approval Page**

I agree to the format and content of this document.

| Approved by: | |
|-----------------------------------------------------------|-------------|
| I Stanley Jankenkun | 28 Oct 2021 |
| Stanley lyadural MD, PhD | Date |
| Vice President, Minical Affairs | |
| Catalyst Pharmaceuticals, Inc. | |
| 355 Alhambra Circle, Suite 1250<br>Coral Gables, FL 33134 | |
| siyadurai@catalystpharma.com | |
| STYLIGHT OF THE THE COST | |
| Authored by: | |
| tal hale | 280ct 2021 |
| Ahmed Belhad, PhD | Date |
| Statistician | |
| STATKING Clinical Services | |
| 759 Wessel Drive | |
| Fairfield, OH 45014 | |
| 513-858-2989 ext. 318 | |
| ahmed@statkingclinical.com | |
| Approved by (internal review): | 9 |
| Muntees | 10 28 2021 |
| lan Lees, MS | Date |
| Statistician | |
| STATKING Clinical Services | |
| 759 Wessel Drive | |
| Fairfield, OH 45014 | |
| 513-858-2989 ext. 327 | |
| ian@statkingclinical.com | |
| Approved by: | |
| Clare Lerger | 16-28-2021 |
| Clare Geiger, RN | Date |
| Project Manager | |
| STATKING Clinical Services | |
| 759 Wessel Drive | |
| Fairfield, OH 45014 | |
| 513-858-2989 ext. 304<br>clare@statkingclinical.com | |
| CIAI CIU/SIAINII II CIII II CAI. CUITI | |

# **Revision History**

N/A

# **Table of Contents**

| 1.0 SYNOPSIS OF STUDY DESIGN PROCEDURES | 6 |
|------------------------------------------------------|----|
| 1.1 Design and Treatment | 6 |
| 1.2 Study Procedures | 7 |
| 1.3 Sample Size | 8 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 8 |
| 2.1 Types of Analyses | 8 |
| 2.2 Analysis Populations | 8 |
| 2.3 Missing Data Conventions | 9 |
| 2.4 Interim Analyses | 9 |
| 2.5 Study Center Considerations in the Data Analysis | 9 |
| 2.6 Documentation and Other Considerations | 9 |
| 3.0 ANALYSIS OF BASELINE SUBJECT CHARACTERISTICS | 9 |
| 4.0 ANALYSIS OF EFFICACY | 10 |
| 4.1 Description of Efficacy Variables | 10 |
| 4.2 Analysis of Efficacy Variables | 10 |
| 5.0 ANALYSIS OF SAFETY | 10 |
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 12 |
| 6.1 Subject Completion | 12 |
| 6.2 Study Drug Administration and Compliance | 12 |
| 6.3 Patient Data Profiles | 12 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 13 |
| 8.0 REFERENCES | 15 |

| APPENDIX A – TABLES, FIGURES | AND LISTING SPECIFICATIONS | 16 |
|------------------------------|----------------------------|----|
| APPENDIX B – TABLE SHELLS | | 18 |

## 1.0 Synopsis of Study Design Procedures

This is an open label observational study. The purpose of this study is to evaluate the long-term safety and tolerability of amifampridine phosphate in patients with muscle-specific receptor tyrosine kinase (MuSK) antibody positive and Acetylcholine receptor (AChR) antibody positive myasthenia gravis (MG) patients who participated in the MSK-002 study. The objectives of this Phase 3 study are as follows:

#### Primary

 To characterize the long-term safety and tolerability of amifampridine phosphate in patients with MG.

#### Secondary

 To assess the clinical efficacy of amifampridine phosphate over time in patients with MG based on change in Myasthenia Gravis Activities of Daily Living Score (MG-ADL).

#### 1.1 Design and Treatment

The study will enroll patients who have completed the MSK-002 study and after all final evaluations for that study have been completed, or those who demonstrated benefit after completing the dose titration period but failed to meet the randomization criteria on Day 0 of MSK-002.

The duration of participation for each patient is expected to be at least 9 months as patients may continue in the study until amifampridine is approved by Regulatory Agencies or the clinical development of amifampridine is terminated for this indication. In addition to amifampridine, patients will continue to receive previous concomitant medications, as needed.

After a new informed consent is signed and inclusion / exclusion criteria for the current protocol are satisfied, eligible patients will be given the optimal dose and dosing schedule that was identified in the Run-in Period from Protocol MSK-002. The findings from the physical exam (including vital signs, weight); 12-lead ECG; clinical laboratory test results (including pregnancy testing) and any ongoing adverse events will be used as the baseline for the Long-Term safety evaluation.

The only efficacy measurement is the MG-ADL which will be completed every 3 or 6 months. Safety and tolerability assessments will be made every 3 or 6 months or more frequently at the discretion of the Investigator. The study will continue until amifampridine is approved by Regulatory Agencies or until development of the product for this indication is halted. The Investigator may alter the dose and dosing frequency during the Long-Term Study as well as schedule additional clinic visits for any reason.

Patients will be seen in the clinic at the end of Months 3, 6, 9, 12, 15, 21, 27, 33, 39. In between the 3-or 6-month visits, patients may also have telephone/video contact with the site, or unscheduled visits, if needed.

### 1.2 Study Procedures

#### Start of Long Term Study

The following procedures are to be performed as scheduled Day 0 and can serve as baseline for the Long-Term study. Any procedure not performed for MSK-002 protocol needs to be completed for this trial.

- Informed Consent for MSK-003;
- o Inclusion/Exclusion criteria for the current study must be verified;
- o Standard 12-lead ECG after 5 minutes in the supine position;
- Complete physical examination including weight;
- Vital signs (seated position), including SBP, DBP, heart rate, respiration, and body temperature;
- Clinical laboratory tests including hematology, chemistry, and urinalysis;
- Urine pregnancy test in females of childbearing potential only;
- o MG-ADL (use data from Day 0 of MSK-002 for all patients);
- Adverse Events (AEs);
- Concomitant medications.

#### • End of Months 3, 6, 9, 12, 15, 21, 27, 33 and 39

The following assessments and procedures will be determined at the end of Months 3, 6, 9, 12, 15 and 21, 27, 33 and 39. Each month has a clinic visit window of ± 1 week. Additional visits are allowed as necessary.

- Assessment of AEs/ Serious Adverse Events (SAEs);
- Complete physical exam with weight;
- Vital signs (seated position), including SBP, DBP, heart rate, respiration, and body temperature;
- Standard 12-lead ECG after 5 minutes in the supine position;
- Clinical laboratory tests including hematology, chemistry, and urinalysis;
- Urine pregnancy test in females of childbearing potential only;
- Concomitant medications;
- IP accountability of medication;
- o MG-ADL.

## End of Study Visit

 Month 39 is the last subject visit in the study, and no IP should be dispensed at Month 39 visit. End of study assessments and procedures listed below should be performed for each subject along

- with final IP accountability. This visit may be incorporated at the scheduled 3-or 6-month visit.
- Assessment of AEs/SAEs;
- Complete physical exam with weight;
- Vital signs (seated position), including SBP, DBP, heart rate, respiration, and body temperature;
- 12-Lead Electrocardiogram (ECG);
- Clinical laboratory tests;
- Urine pregnancy test in females of childbearing potential only;
- Concomitant medications;
- MG-ADL.

#### 1.3 Sample Size

The study is not powered with respect to any endpoint but is an observational study to assess long term safety and lack of tolerance to the effects of amifampridine on MG-ADL.

## 2.0 Data Analysis Considerations

#### 2.1 Types of Analyses

The following standards will be applied for the analyses unless otherwise specified. Simple summary statistics (descriptive statistics) for continuous data are: n (number of non-missing observations), mean, median, standard deviation, minimum, and maximum. The frequency count and percentage will be used to summarize categorical data. Summary statistics will be presented by treatment. All data collected will be presented in the by-subject data listings, sorted by subject and by time point, where appropriate.

#### 2.2 Analysis Populations

The following analysis populations will be defined:

**Safety Population:** The safety population will consist of all subjects who are enrolled in the study and have received at least one dose of amifampridine.

**Full Analysis Set (FAS), Intent to Treat Population:** This population consists of all subjects who receive at least 1 dose of IP (amifampridine) and have at least one post-treatment efficacy assessment.

The FAS population will be the primary data set for all effectiveness analyses. The Safety population will be used to analyze all safety variables and baseline characteristics.

#### 2.2.1 Subgroup Definitions

Subgroup analyses for safety will be performed independently on the MuSK-MG and AChR-MG groups. No pooled analyses are planned.

### 2.3 Missing Data Conventions

No missing value imputation will be used. That is, all analyses will be based on the observed data (i.e., complete case analysis).

#### 2.4 Interim Analyses

There are no interim analyses planned for this study.

#### 2.5 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI).

There will be no selective pooling of study centers in the analysis. All calculations will be made on the combined results of all centers.

#### 2.6 Documentation and Other Considerations

The data analyses will be conducted using SAS® Software, version 9.4 or later.

All SAS code used to generate SDTM and ADaM datasets and the final tables and listings will be provided.

# 3.0 Analysis of Baseline Subject Characteristics

Baseline and demographic characteristics will be summarized by MG type and overall for all subjects in the safety population. Age and baseline height and weight will be displayed via summary statistics (mean, median, sample size, standard deviation, minimum, and maximum). Gender and ethnicity will be summarized via counts and percentages.

A detailed listing of demographics data for each subject will also be provided as shown in Appendix B.

## 4.0 Analysis of Efficacy

### 4.1 Description of Efficacy Variables

For this study the efficacy endpoints are secondary endpoints. The efficacy variable is the MG-ADL score at months 3, 6, 9, 12, 15, 21, 27, 33 and 39.

#### 4.2 Analysis of Efficacy Variables

#### 4.2.1 Secondary Efficacy Analysis

Summary statistics (n, mean, standard deviation, minimum, median and maximum) for the MG-ADL score at Months 3, 6, 9, 12, 15, 21, 27, 33 39, and change from baseline (Day 0 of MSK-002 for all patients) will be presented

All secondary efficacy data will be listed as shown in Appendix B.

## 5.0 Analysis of Safety

For this study, the primary endpoint is safety and tolerability of amifampridine at Months 3, 6, 9, 12, 15 and 21, 27, 33 and 39.

The safety variables for this study are:

- AEs
- Vital signs
- Physical examination
- ECG
- Clinical laboratory results
- Concomitant medications

#### Adverse Events

All AEs will be observed for each subject from enrollment until termination from the study. Prior to analysis, all AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA). Based on these coded terms, treatment emergent AEs (TEAEs) will be summarized using system organ class and preferred term by MG type and overall for all subjects in the safety population. This analysis will be repeated for serious TEAEs (TESAEs).

TEAEs will also be summarized by severity and relationship to IP. An overall summary table will provide the highest relationship and maximum severity observed per subject, as well as the counts of subjects with at least one TESAE.

All AEs will be listed, regardless of whether or not they were treatment emergent.

#### **Vital Signs**

Summary statistics (mean, median, sample size, standard deviation, minimum, and maximum) will be computed on the raw and change from baseline values for each vital sign parameter by time point, for each MG type. The screening time point will serve as baseline. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

#### **Physical Exam**

A shift table of physical exam results will be created showing the shifts in results by parameter relative to the normal ranges. The number and percentage of subjects with the following shifts will be presented: normal/normal, normal/low, normal/high, low/low, low/normal, low/high, high/low, high/normal, and high/high. The physical exam data collected at screening, or termination from the study will be listed.

#### Electrocardiogram

A table containing descriptive statistics for QTc values measured at screening, or termination from the study and CFB by MG type will be created. A shift table showing normal/normal, normal/abnormal, abnormal/normal and abnormal/abnormal shifts as counts and percentages will be created. The ECG data collected will be listed.

#### **Clinical Laboratory Results**

Tables containing descriptive statistics for serum chemistry, hematology and urinalysis values measured at screening (pre-treatment level, the baseline value), or termination from the study and Change From Screen Level (CFS) by MG type will be created. In addition, a shift table will be constructed to show the shifts in laboratory results by parameter relative to the normal ranges. The number and percentage of subjects with the following shifts will be presented: normal/normal, normal/low, normal/high, low/low, low/normal, low/high, high/low, high/normal, and high/high.

#### **Concomitant Medications**

A table of the WHO-coded medications will be constructed by MG type group and overall with medications summarized by anatomical therapeutic chemical (ATC) level 3 term and preferred term. The number and percent of subjects on each drug will be summarized. A data listing for all concomitant medications will be provided.

# 6.0 Other Relevant Data Analyses/Summaries

#### 6.1 Subject Completion

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of the number of subjects withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table will include summary counts and percentages by MG type. A data listing of all subject completion and withdrawal data will also be constructed.

#### **6.2 Study Drug Administration and Compliance**

Duration of treatment administration will be computed per subject as:

Duration (in days) = (Date of last dose) – (Date of randomization) + 1

Duration will be summarized using descriptive statistics by treatment group.

Compliance will be computed per subject as:

Compliance = 100%\*(Number consumed)/(Number prescribed),

where number prescribed is defined as the duration times the number of tablets to have been taken daily. Compliance will be summarized using descriptive statistics by MG type.

#### 6.3 Patient Data Profiles

A Patient Data Profile listing will be provided. It will contain demographic information, randomization information, all endpoint assessments and laboratory measurements. See Appendix B, Data Listing 18 for full details. Some variation in the appearance of this table is acceptable to accommodate unformatted SAS® output provided that all information is present.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in Appendix B |
|---|---|---|---|
| 1 | Subject Disposition (All subjects) | X | X |
| 2 | Demographics and Baseline Data Summary Statistics – Continuous Variables (Safety Population) | Х | X |
| 3 | Demographics and Baseline Data Summary Statistics – Categorical Variables (Safety Population) | X | Х |
| 4 | Summary of Study Drug Administration and Compliance (Safety Population) | X | Х |
| 5 | MG-ADL Total Score Summary Statistics by Time Point and MG Type (FAS Population) | Х | Х |
| 6 | Number and Percent of Subjects with Treatment<br>Emergent Adverse Events (Safety Population) | Х | Х |
| 7 | Summary of Treatment Emergent Adverse Events (Safety Population) | Х | Х |
| 8 | Number and Percent of Subjects with Treatment Emergent Serious Adverse Events (Safety Population) | Х | Х |
| 9 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to MG Type (Safety Population) | Х | Х |
| 10 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade (Safety Population) | Х | Х |
| 11 | ECG Shift Summary Statistics by MG Type (Safety Population) | Х | Х |
| 12 | ECG QTc Interval Summary Statistics by Time Point and MG Type (Safety Population) | Х | Х |
| 13 | Serum Chemistry Clinical Laboratory Summary<br>Statistics by Time Point and MG Type (Safety<br>Population) | х | Х |
| 14 | Hematology Clinical Laboratory Summary Statistics by Time Point and MG Type (Safety Population) | Х | |
| 15 | Urinalysis Clinical Laboratory Summary Statistics by Time Point and MG Type (Safety Population) | Х | |
| 16 | Serum Chemistry Shift Table by MG Type (Safety Population) | х | Х |
| 17 | Hematology Shift Table by MG Type (Safety Population) | Х | |
| 18 | Urinalysis Shift Table by MG Type (Safety Population) | Х | |
| 19 | Vital Sign Parameters Summary Statistics by MG Type (Safety Population) | х | Х |
| 20 | Vital Signs Shift Table by MG Type (Safety Population) | Х | X |
| 21 | Number and Percent of Subjects Taking Concomitant Medications by ATC Level 3 and Preferred Term (Safety Population) | х | Х |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | X | X |
| DL2 | Protocol Deviations Data Listing | X | X |
| DL3 | Demographics Data Listing | X | X |
| DL4 | Subjects Excluded from FAS Population Data Listing | X | X |
| DL5 | Subjects Excluded from PP Population Data Listing | X | Х |
| DL6 | Medical History Data Listing | X | Х |
| DL7 | Prior and Concomitant Medications Data Listing | X | Х |
| DL8 | Adverse Events Data Listing | X | Х |
| DL9 | Physical Exam Data Listing | X | Х |
| DL10 | Vital Signs Data Listing | X | X |
| DL11 | ECG Data Listing | X | Х |
| DL12 | Study Drug Administration Data Listing | X | Х |
| DL13 | Serum Chemistry Data Listing | X | Х |
| DL14 | Hematology Data Listing | X | Х |
| DL15 | Urinalysis Data Listing | Х | Х |
| DL16 | Amifampridine Level Data Listing | X | Х |
| DL17 | MG-Activities of Daily Living Data Listing | Х | Х |
| DL18 | Subject Data Profile | X | X |

# 8.0 References

NA

## Appendix A - Tables, Figures and Listing Specifications

#### Orientation

Tables, figures, and listings will be displayed in landscape with the exception of the Patient Data Profile Listing (DL18), which will be in portrait layout.

#### **Margins**

Margins will be 1 inch on all sides. Table, figure, and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### **Headers**

The table number will be on the second line of the title area. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, one line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (Date)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this Statistical Analysis Plan (SAP) will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

#### **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

### **Computation Values for Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (e.g., for a missing day value, the value displayed is in mmm-yyyy format). When date computations are necessary, the following table indicates the substitutions used in order to make those computations.

| Scenario | Value Used for Computations |
|---|---|
| Start date – Missing month and day values | January 1 of the indicated year |
| Start date – Missing day values | The first day of the indicated month |
| Stop date – Missing month and day values | December 31 of the indicated year |
| Stop date – Missing day values | The last day of the indicated month |

# Appendix B – Table Shells

Page x of y

Table 1. Subject Disposition (All subjects)
Catalyst Pharmaceuticals, Inc. - MSK-003

| | | | MuSK | | AChR | 70 | verall |
|---|---|---|---|---|---|---|---|
| Screen Failures | | | | | | | XX |
| Enrolled | | | xx | | XX | | xx |
| Completed | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| Withdrawn | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| Reason for Withdrawal | Adverse Event Lost To Follow-Up Death Physician Decision Protocol Deviation Study Terminated by Sponsor Withdrawal by Subject Other | xx<br>xx<br>xx<br>xx<br>xx<br>xx | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) | XX<br>XX<br>XX<br>XX | (xxx%) | XX<br>XX<br>XX<br>XX<br>XX | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) |

The denominator for all percentages in the table is the number of enrolled subjects in the respective MG treatment group and overall. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics - Continuous Variables Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Variable | MG Type | Mean | Std Dev | n | Min | Max | Median |
|----------------------|---------|------|---------|-----|-----|-----|--------|
| Age (years) | MuSK | XXX | XXX | XXX | XXX | XXX | XXX |
| | AChR | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline Weight (kg) | MuSK | XXX | xxx | XXX | xxx | XXX | xxx |
| | AChR | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline Height (cm) | MuSK | XXX | xxx | XXX | xxx | XXX | XXX |
| | AChR | xxx | XXX | XXX | XXX | XXX | XXX |
| | Overall | xxx | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics - Categorical Variables

Catalyst Pharmaceuticals, Inc. - MSK-003

Safety Population (N=xxx)

| Demographics<br>Variable | Category | MuSK<br>(N=xxx) | AChR<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|---|
| Gender | Male | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Female | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Ethnicity | Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Not Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 4. Summary of Study Drug Administration and Compliance Catalyst Pharmaceuticals, Inc. - MSK-003
Safety Population (N=xxx)

| | | MuSK | AChR |
|-----------------|------------------|-----------|-----------|
| | Statistic | (N=xxx) | (N=xxx) |
| Duration (days) | n | XXX | XXX |
| | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | Median | xxx | XXX |
| | Minimum, Maximum | xxx, xxx | xxx, xxx |
| Compliance (%) | n | xxx | xxx |
| | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | Median | xxx | xxx |
| | Minimum, Maximum | xxx. xxx | xxx. xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 5. MG-ADL Total Score Summary Statistics by Time Point and MG Type Catalyst Pharmaceuticals, Inc. - MSK-003  $FAS \ \ Population \ \ (N=xxx)$ 

Part 1 of 2

| MG Type <sup>a</sup> | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Std<br>Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|
| MuSK | Day 0 of MSK-002<br>(Baseline) | RAW | XXX | xxx | xxx | XXX | XXX | xxx |
| | Month 3 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 6 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 9 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 12 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 15 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 21 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 27 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 33 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 39 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> The treatment of MG result will be the result obtained at Months 3, 6, 9, 12, 15, 21, 27, 33 and 39, unless the subject discontinued treatment of MG early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 5. MG-ADL Total Score Summary Statistics by Time Point and MG Type Catalyst Pharmaceuticals, Inc. - MSK-003 FAS Population (N=xxx)

Part 2 of 2

| MG Type <sup>a</sup> | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Std<br>Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|
| AChR | Day 0 of MSK-002<br>(Baseline) | RAW | xxx | xxx | XXX | xxx | xxx | XXX |
| | Month 3 | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 6 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 9 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 12 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 15 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 21 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 27 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 33 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 39 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> The treatment of MG result will be the result obtained at Months 3, 6, 9, 12, 15, 21, 27, 33 and 39, unless the subject discontinued treatment of MG early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline.

Page x of y

Table 6. Number and Percent of Subjects with Treatment Emergent Adverse Events
Catalyst Pharmaceuticals, Inc. - MSK-003
Safety Population (N=xxx)

| Adverse Event Category*: | MuSK<br>(N=xxx) | AChR<br>(N=xxx) |
|---|---|---|
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 7. Summary of Treatment Emergent Adverse Events Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxxx)

| | MuSK<br>(N=xxx) | AChR<br>(N=xxx) |
|---|---|---|
| Subjects with at Least One Treatment Emergent Adverse Event (TEAE) | xxx (xxx%) | xxx (xxx%) |
| Maximum TEAE Severity Grade | | |
| Mild (Grade 1) | xxx (xxx%) | xxx (xxx%) |
| Moderate (Grade 2) | xxx (xxx%) | xxx (xxx%) |
| Severe (Grade 3) | xxx (xxx%) | xxx (xxx%) |
| Life-threatening (Grade 4) | xxx (xxx%) | xxx (xxx%) |
| Death (Grade 5) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Treatment | | |
| Not Related | xxx (xxx%) | xxx (xxx%) |
| Possibly | xxx (xxx%) | xxx (xxx%) |
| Probably | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One Serious TEAE | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 8. Number and Percent of Subjects with Treatment Emergent Serious Adverse Events Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Adverse Event Category*: | MuSK<br>N=xxx) | AChR<br>(N=xxx) |
|---|---|---|
| Total Number of Serious Treatment Emergent<br>Adverse Events (TESAEs) | xxx | xxx |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 9. Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to MG Type

Catalyst Pharmaceuticals, Inc. - MSK-003

Safety Population (N=xxx)

MuSK AChR (N=xxx)(N=xxx)Adverse Event Categorya: Not Related Possibly Probably Not Related Possibly Probably Total Number of Treatment Emergent Adverse XXX XXX XXX XXX XXX XXX Events (TEAEs) Subjects with at Least One TEAE xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 1 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) Preferred Term 1 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) Preferred Term 2 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) System Organ Class 2 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) Preferred Term 1 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) Preferred Term 2 xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%)

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 10. Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade
Catalyst Pharmaceuticals, Inc. - MSK-003
Safety Population (N=xxx)

Part 1 of 2

MuSK

| | (N=XXX) | | | | |
|---|---|---|---|---|---|
| Adverse Event Categorya: | Grade 1 Grade 2 Grade 3 | | Grade 4 | Grade 5 | |
| Total Number of Treatment Emergent<br>Adverse Events (TEAEs) | xxx | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | , , | , , | , , | xxx (xxx%) | , , |
| Preferred Term 1 Preferred Term 2 | , , | , , | , , | xxx (xxx%) | , , |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 10. Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

Part 2 of 2

AChR

| | (N=xxx) | | | | |
|---|---|---|---|---|---|
| Adverse Event Categorya: | Grade 1 Grade 2 | | Grade 3 | Grade 4 | Grade 5 |
| Total Number of Treatment Emergent<br>Adverse Events (TEAEs) | xxx | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | , , | , , | , , | xxx (xxx%) | , , |
| Preferred Term 1 Preferred Term 2 | , , | , , | , , | xxx (xxx%) | , , |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 11. ECG Shift Summary Statistics by MG Type Catalyst Pharmaceuticals, Inc. MuSK-003 Safety Population (N=xxx)

| MG Type | Screening (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Normal | Screening (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Abnormal | Screening (Baseline) Abnormal/ End of Study <sup>a</sup> Normal | Screening (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Abnormal |
|---|---|---|---|---|
| MuSK (N=xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| AChR (N=xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (month day, year)

<sup>&</sup>lt;sup>a</sup> End of study is at least 9 months (i.e. until amifampridine is approved by Regulatory Agencies for the treatment of MG or the development program is discontinued for this indication).

Page x of y

Table 12. ECG QTc Interval Summary Statistics
By Time Point and MG Type
Catalyst Pharmaceuticals, Inc. MuSK-003
Safety Population (N=xxx)

Part 1 of 2

| | | Data | | Mean | Std | | | |
|---|---|---|---|---|---|---|---|---|
| MG Type | Visit | Typeª | n | (msec) | Dev | Min | Median | Max |
| MuSK | Screening (Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | xxx |
| | Month 3 | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 6 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 9 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 12 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 15 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 21 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 27 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 33 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 39 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | xxx |

STATKING Clinical Services (month day, year)

 $<sup>^{\</sup>mathrm{a}}$  CFB refers to Change from Baseline (Screening ECG).

Page x of y

Table 19. ECG QTc Interval Summary Statistics
By Time Point and MG Type
Catalyst Pharmaceuticals, Inc. MuSK-003
Safety Population (N=xxx)

Part 2 of 2

| | | Data | | Mean | Std | | | |
|---|---|---|---|---|---|---|---|---|
| MG Type | Visit | Typeª | n | (msec) | Dev | Min | Median | Max |
| AChR | Screening (Baseline) | RAW | XXX | xxx | XXX | xxx | xxx | XXX |
| | Month 3 | RAW | xxx | xxx | XXX | xxx | xxx | xxx |
| | | CFB | XXX | xxx | XXX | XXX | XXX | xxx |
| | Month 6 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 9 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 12 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 15 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 21 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 27 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 33 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Month 39 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (month day, year)

 $<sup>^{\</sup>rm a}$  CFB refers to Change from Baseline (Screening ECG).

Page x of y

Table 13. Serum Chemistry Clinical Laboratory Summary Statistics by Time Point and MG Type Catalyst Pharmaceuticals, Inc. MuSK-003 Safety Population (N=xxx)

Laboratory Panel: Serum Chemistry

| Parameter | MG Type | Visit | Data | | | Std | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Typeª | n | Mean | Dev | Min | Median | Max |
| xxxxxxxxxxxxxxx | MuSK | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | XXX | xxx |
| | | End of study | RAW | xxx | XXX | XXX | xxx | xxx | xxx |
| | | - | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| xxxxxxxxxxxxxxx | AChR | Screening (Baseline) | RAW | xxx | XXX | xxx | xxx | xxx | xxx |
| | | End of study | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | _ | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Source Listing: Data Listing 13

The format of this table is repeated for hematology and urinalysis panels.

<sup>&</sup>lt;sup>a</sup> CFB refers to Change from Baseline (Screening sample).

Page x of y

Table 16. Serum Chemistry Shift Table by MG Type Catalyst Pharmaceuticals, Inc. MSK-003 Safety Population (N=xxx)

| Lab Parameter | MG Type | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxxx | MuSK | (xxx%) | xxx<br>(xxx%) | (xxx%) | (xxx%) | (xxx%) | xxx<br>(xxx%) | (xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) |
| xxxxxxxx | AChR | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) |

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas Source Listing: Data Listing 13

## Table repeats for hematology and urinalysis panels.

<sup>&</sup>lt;sup>a</sup> Shifts represent screening/end of study, where end of study is least 9 months (i.e. until amifampridine is approved by Regulatory Agencies for the treatment of MG or the development program is discontinued for this indication).
Page x of y

Table 19. Vital Signs Parameters Summary Statistics by MG Type Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

Part 1 of 2

| | | | | | | | Std | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Vital Sign Paramet | ter (units) MG | Type Visit | Da | ta Typeª | n | Mean | Dev | Min | Max N | Median |
| xxxxxxxxxx (xxx) | MuS | SK Screeni | ng (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | D. 7. 7. | | | | | | |
| | | Month 3 | i | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 6 | | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 9 | ı | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | xxx | XXX | XXX |
| | | Month 1 | 2 | RAW | XXX | XXX | XXX | XXX | xxx | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | xxx | XXX |
| | | Month 1 | 5 | RAW | xxx | XXX | XXX | XXX | XXX | xxx |
| | | | | CFB | XXX | XXX | XXX | XXX | xxx | xxx |
| | | Month 2 | 1 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 2 | 7 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 3 | 3 | RAW | XXX | XXX | XXX | xxx | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | xxx | xxx |
| | | Month 3 | 9 | RAW | XXX | XXX | XXX | XXX | xxx | xxx |
| | | | | CFB | xxx | | | | XXX | xxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> RAW = observed data recorded in database; CFB = change from baseline

Page x of y

Table 19. Vital Signs Parameters Summary Statistics by MG Type Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

Part 2 of 2

| | | | | | | Std | | | |
|---|---|---|---|---|---|---|---|---|---|
| Vital Sign Parameter (units) | MG Type | Visit | Data Typeª | n | Mean | Dev | Min | Max | Median |
| xxxxxxxxx (xxx) | AChR | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 3 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 6 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 9 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 12 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 15 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 21 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 27 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 33 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Month 39 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> RAW = observed data recorded in database; CFB = change from baseline

Page x of y

## Table 20. Vital Signs Shift Table by MG Type Catalyst Pharmaceuticals, Inc. MSK-003 Safety Population (N=xxx)

| Lab Parameter | MG Type <sup>a</sup> | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxxxx | MuSK | xxx<br>(xxx%) | xxx<br>(xxx%) | (xxx%) | xxx<br>(xxx%) | (xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx (xxx%) |
| xxxxxxxxx | AChR | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> End of study is least 9 months (i.e. until amifampridine is approved by Regulatory Agencies for the treatment of MG or the development program is discontinued for this indication). withdrawal from study, whichever is earlier.

STATKING Clinical Services (month day, year)

Page x of y

Table 21. Number and Percent of Subjects Taking Concomitant Medications by ATC Level 3 and Preferred Term

Catalyst Pharmaceuticals, Inc. - MSK-003

Safety Population (N=xxx)

| Concomitant Medication Category <sup>a,b</sup> | Musk<br>(N=xxx) | AChR<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| ATC Level 3 Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term WHO Preferred Term | xxxx (xxxx%)<br>xxxx (xxxx%) | xxxx (xxxx%)<br>xxxx (xxxx%) | xxxx (xxxx%)<br>xxxx (xxxx%) |
| | , , | , , | , |
| ATC Level 3 Term WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) xxxx (xxxx%) | xxxx (xxxx%)<br>xxxx (xxxx%) |

a Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxx.

b Concomitant medication categories will include anatomical therapeutic chemical (ATC) level 3 term followed by preferred term. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

## Data Listing 1. Subject Disposition Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003

| Subject | | | | |
|---|---|---|---|---|
| No. | MG Type | Disposition Status | Date of Disposition | Withdrawal Reason |
| XXXX | xxxxxx | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx |
| XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXX | xxxxxx | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxx |
| XXXX | xxxxxx | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 2. Protocol Deviations Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Subject | | Date of | | Deviation Major or |
|---|---|---|---|---|
| No. | MG Type | Deviation | Deviation Description | Minor |
| XXXX | XXXXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXX | XXXXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXX | XXXXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXX | XXXXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 3. Demographics Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| | | Informed | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | Consent | Date of | Age | | | Screening | |
| MG Type | No. | Date | Birth | (yrs) | Gender | Ethnicity | Weight (kg) | Height (cm) |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| YYYYYY | YYYY | XXXXXX | ×××××× | XXX | XXXXXX | XXXXXX | ×××××× | XXXXXX |

 ${\tt STATKING~Clinical~Services~(DD-MMM-YYYY)}$ 

Page x of y

Data Listing 4. Subjects Excluded from FAS Population Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003
Safety Population (N=xxx)

| MG Type | Subject No. | Reason for Exclusion |
|---------|-------------|----------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |

 ${\tt STATKING~Clinical~Services~(DD-MMM-YYYY)}$ 

Page x of y

Data Listing 5. Subjects Excluded from PP Population Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003

All Enrolled Subjects (N=xxx)

| MG Type | Subject No. | Reason for Exclusion |
|---------|-------------|----------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 6. Medical History Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

MedDRA System Organ Classa/

| MG Type | Subject<br>No. | MedDRA Preferred Term/<br>CRF Verbatim Term | Start Date | Ongoing? |
|---|---|---|---|---|
| xxxxxx | xxxx | ******** | xxxxxxx | xxx |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxx | XXX |

<sup>&</sup>lt;sup>a</sup> Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 7. Prior and Concomitant Medications Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

WHO Preferred Terma/

| W0 T | Subject | Verbatim Drug Name/<br>Indication/<br>ATC Level 1 Term/ | Start | Stop | | |
|---|---|---|---|---|---|---|
| MG Type | No. | ATC Level 3 Term | Date | Date | Route | Ongoing? |
| xxxxxx | xxxxxxx | ************************************** | xxxxxx | xxxxxx | xxxxx | xxxxx |
| xxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxx | xxxxxx | xxxxx | xxxxx |

 $<sup>^{\</sup>rm a}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 8. Adverse Events Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| | | Start<br>Date and<br>Time/ | | MedDRA System<br>Organ Class <sup>a</sup> /<br>MedDRA Preferred | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | End Date | Treatment | Term/ | Severity | Relation to | | |
| MG Type | No. | and Time | Start Date | CRF Verbatim Term | Grade | Treatment | Serious? | Outcome |
| xxxxxx | xxxxxxxx | xxxxxx | xxxxxxx | xxxxxxxxxxxxxx | xxxxxxx | xxxxxxx | XXX | xxxxxxx |
| | | xxxxxxx/ | XXXXXXX | XXXXXXXXXXXXXXXX | | | | |
| | | XXXXXXX | | XXXXXXXXXXXXXXXX | | | | |
| | | xxxxxx | | | | | | |
| XXXXXX | xxxxxxxx | xxxxxx | xxxxxx | xxxxxxxxxxxxxxx | xxxxxxx | xxxxxxxx | xxx | xxxxxxx |
| | | xxxxxxx/ | XXXXXXX | xxxxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | xxxxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | | | | | |

 $<sup>^{\</sup>rm a}$  Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 9. Physical Exam Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| | Subject | | Date | | | |
|---|---|---|---|---|---|---|
| MG Type | No. | Visit | Conducted | Body System | Result | Abnormality |
| - | | | | | | |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | XXXXXXX | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxx | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 10. Vital Signs Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| MG Type | Subject<br>No. | Visit | Date | Time | Temp. | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Heart<br>Rate<br>(bpm) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxx | xxx | XXX | xxx |
| | | | | xxxxx | xxx | xxx | xxx | xxx |
| | | | | XXXXX | XXX | XXX | XXX | XXX |
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | XXX | xxx | XXX | xxx |
| | | | | XXXXX | XXX | XXX | xxx | XXX |
| | | | | XXXXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 11. ECG Data Listing Catalyst Pharmaceuticals - MuSK-003 Safety Population (N=xxx)

| | Subject | | | | | Heart | PR | QRS | QT | ECG Assessment/ If |
|---|---|---|---|---|---|---|---|---|---|---|
| MG Type | No. | Age | Time Point | Date | Time | Rate | Interval | Duration | Interval | Abnormal, Specify |
| XXXX | XXXXXX | XXXX | Screen | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | xxxxxxxxxxxxxxx |
| | | | Month 3 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | xxxxxxxxxxxxxxx |
| | | | Month 9 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | xxxxxxxxxxxxxxx |
| | | | Month 12 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | XXXXXXXXXXXXXXXXX |
| | | | Month 15 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | xxxxxxxxxxxxxxx |
| | | | Month 21 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | XXXXXXXXXXXXXXXXX |
| | | | Month 27 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | XXXXXXXXXXXXXXXXX |
| | | | Month 33 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | XXXXXXXXXXXXXXXX |
| | | | Month 36 | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | | | | XXXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Study Drug Administration Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| MG Type | Subject<br>No. | Treatment<br>Start<br>Date | Treatment<br>End Date | Treatment<br>Duration<br>(Days) | Tablets<br>Consumed | Dose (mg/day) | Tablets<br>Prescribed <sup>a</sup> | Compliance (%)b |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxx | XXXXXX | XXX | xxx | xxx | xxx | xxx |
| xxxxxx | xxxx | xxxxxx | xxxxxx | xxx | xxx | XXX | xxx | XXX |

 ${\tt STATKING~Clinical~Services~(DD-MMM-YYYY)}$ 

<sup>&</sup>lt;sup>a</sup> Number of tablets prescribed is computed as the duration times the number of tablets to have been taken daily.

b Compliance is computed as 100%\*(number of tablets consumed)/(number of tables prescribed).

Page x of y

Data Listing 13. Serum Chemistry Data Listing Catalyst Pharmaceuticals - MuSK-003 Safety Population (N=xxx)

| | | | | Parameter | | Assessment/ If Abnormal, |
|---|---|---|---|---|---|---|
| MG Type | Subject No. | Time Point | Date | (Units) | Value | Specify |
| | | | | | | _ |
| XXXX | XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX | xxxxxx/ |
| | | | | | | xxxxxxxxxxxxxxx |
| | | | | XXXXX | XXXXX | xxxxxx/ |
| | | | | | | XXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 14. Hematology Data Listing Catalyst Pharmaceuticals - MuSK-003 Safety Population (N=xxx)

| | | | | P | arameter | A | Assessment/ If Abnormal, |
|---|---|---|---|---|---|---|---|
| 1 | MG Type | Subject No. | Time Point | Date | (Units) | Value | Specify |
| | XXXX | XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | xxxxxxxxxxxxxxx |
| | | | | | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | xxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 15. Urinalysis Data Listing Catalyst Pharmaceuticals - MuSK-003 Safety Population (N=xxx)

| | | | | P | arameter | A | Assessment/ If Abnormal, |
|---|---|---|---|---|---|---|---|
| 1 | MG Type | Subject No. | Time Point | Date | (Units) | Value | Specify |
| | XXXX | XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | xxxxxxxxxxxxxxx |
| | | | | | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | | | xxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 16. Amifampridine Levels Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| | | Subject | | Date of | Time of | Amifampridine Level |
|---|---------|---------|----------|---------|---------|---------------------|
| | MG Type | No. | Visit | Sample | Sample | (Units) |
| - | xxxxxx | xxxx | xxxxxxx | xxxxxxx | xx:xx | xxxxxxxxxxxxxxxxx |
| | xxxxxx | xxxx | xxxxxxxx | xxxxxxx | xx:xx | xxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

## Data Listing 17. MG-Activities of Daily Living Data Listing Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| | Subject | | | | Change from | Best-Case Imputed | Worst-Case |
|---|---|---|---|---|---|---|---|
| MG Type | No. | Visit | ADL Score | Baseline Value | Baseline | Value | Imputed Value |
| xxxxx | xxxx | xxxxxxx | xxxx | xxxx | xxxx | xxxx | xxxx |
| XXXXXX | xxxx | xxxxxxx | XXXX | xxxx | XXXX | xxxx | xxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 18. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Study Numbe | er: MSK-003 | Site: xxxxxxxxx | Subject ID: xxxxx | |
|---|---|---|---|---|
| Age (yrs): | ion Code: xxxx<br>xxxx<br>Weight (kg): xxxx | Treatment: xxxxxx Gender: xxxxxx MG Type: xxxxxxx | Dose: xxxxxx<br>Ethnicity: xxxxxxx | Dose Group: xxxx |
| Endpoint Me | easurements | | | |
| Myasthenia | Gravis - Activities | of Daily Living Scores | | |
| Visit | Dat | e | Score | CFB |
| Baseline | xx- | xxx-xxxxx Total | XXXXX | |
| Month x | XX- | xxx-xxxx Total | xxxxx | XXXXX |
| Ouantitativ | ve Myasthenia Gravis | Scores | | |
| Visit | Date | Item | Score | CFB |
| Baseline | xx-xxx-xxxx | Double Vision Sec. | xxxxx | |
| | | Bothersome Ptosis | xxxxx | |
| | | Facial Muscles | xxxxx | |
| | | Swallowing | XXXXX | |
| | | Speech Following Counting From 1-50 | XXXXX | |
| | | Right Arm Outstretched | XXXXX | |
| | | Left Arm Outstretched | xxxxx | |
| | | Forced Vital Capacity | xxxxx | |
| | | Right Hand Grip (kg) | XXXXX | |
| | | Left Hand Grip (kg) | xxxxx | |
| | | Head, Lifted | xxxxx | |
| | | Right Leg Outstretched | xxxxx | |
| | | Left Leg Outstretched | XXXXX | |
| | | Limb Total | XXXXX | |
| | | Total | XXXXX | |
| Month x | xx-xxx-xxxx | Double Vision Sec. | XXXXX | XXXXX |
| | | Bothersome Ptosis | XXXXX | XXXXX |
| | | Facial Muscles | XXXXX | XXXXX |
| | | Swallowing | XXXXX | XXXXX |
| | | Speech Following Counting From 1-50 | XXXXX | XXXXX |
| | | Right Arm Outstretched | XXXXX | XXXXX |
| | | Left Arm Outstretched | XXXXX | XXXXX |
| | | Forced Vital Capacity | XXXXX | XXXXX |
| | | Right Hand Grip (kg) | XXXXX | XXXXX |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

STATKING Clinical Services (DD-MMM-YYYY)

 $<sup>^{\</sup>rm b}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxx.

Page x of y

Data Listing 18. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Study Number: | | Site: xxxxxxxxx | Subject ID: | XXXXX | |
|---|---|---|---|---|---|
| | Myasthenia Gravis Sco | ores | | | |
| Visit | Date | Item | | Score | CF |
| Month x | XX-XXX-XXXXX | Left Hand Grip (kg) | | XXXXX | XXXX |
| | | Head, Lifted | | XXXXX | XXXX |
| | | Right Leg Outstretched | | XXXXX | XXXX |
| | | Limb Total | | XXXXX | XXXX |
| | | Total | | XXXXX | XXXX |
| Safety Measur | rements | | | | |
| Laboratory Va | | | | | |
| Visit | Date | Parameter (units) | Result | Abnormal Criterion | |
| Baseline | xx-xxx-xxx | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | XXXX | | |
| Electrocardio | ogram Values | | | | |
| Visit | Date | Parameter (units) | Result | Abnormal Criterion | |
| Baseline | xx-xxx-xxx | xxxxxxxxxxxxxxxx | XXXX | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | xxxxxxxxxxxxxxxx | xxxx | | |
| | | XXXXXXXXXXXXXXXXXX | XXXX | | |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX | | |
| Month x | xx-xxx-xxx | | | | |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXX | | |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxx<br>xxxx | | |
| | | ************************************** | xxxx<br>xxxx<br>xxxx | | |
| Month x Vital Sign Va | | ************************************** | xxxx<br>xxxx<br>xxxx | Abnormal Criterion | |
| Vital Sign V <i>a</i><br>Visit | alues | ************************************** | xxxx<br>xxxx<br>xxxx<br>xxxx | Abnormal Criterion | |
| Vital Sign Va | alues<br>Date | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxx<br>xxxx<br>xxxx<br>xxxx<br>Result | Abnormal Criterion | |
| Vital Sign V <i>a</i><br>Visit | alues<br>Date | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxx<br>xxxx<br>xxxx<br>xxxx<br>Result<br>xxxx | Abnormal Criterion | |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

STATKING Clinical Services (DD-MMM-YYYY)

 $<sup>^{\</sup>rm b}$  Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxxx.

Page x of y

Data Listing 18. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-003 Safety Population (N=xxx)

| Study Number: MS | K-003 | Site: xxxxxxx | Site: xxxxxxxxx | | XXXX |
|---|---|---|---|---|---|
| | · | · | | · | |
| Vital Sign Value | g. | | | | |
| Visit | Date | Parameter (units) | ) | Result | Abnormal Criterion |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXX | XXXX | |
| | | xxxxxxxxxxxxxxx | XXXX | xxxx | |
| | | xxxxxxxxxxxxxxxx | XXXX | xxxx | |
| | | xxxxxxxxxxxxxxx | XXXX | xxxx | |
| Month x | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXX | xxxx | |
| | | xxxxxxxxxxxxxxx | XXXX | xxxx | |
| | | XXXXXXXXXXXXXXXX | XXXX | xxxx | |
| | | xxxxxxxxxxxxxx | XXXX | XXXX | |
| Adverse Events | | | | | |
| Preferred Term | Date | System Organ Clas | SS | Severity | Treatment Related? |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXXX | xxxx | |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXXX | xxxx | xxxxxxxxxx |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXXX | xxxx | xxxxxxxxxx |
| xxxxxxxxx | XX-XXX-XXXX | xxxxxxxxxxxxxx | XXXXX | XXXX | XXXXXXXXXX |
| Concomitant Medi | cations | | | | |
| Preferred Term | Dose (units, freq) | Start Date | Stop Date | | |
| XXXXXXX | xxxxx (xxxx, xxxx) | xx-xxx-xxxx | xx-xxx-xxxx | | |
| | | xx-xxx-xxxx | xx-xxx-xxxx | | |
| XXXXXX | xxxxx (xxxx, xxxx) | AX-XXX-XXXX | 2121 212121 21212121 | | |
| XXXXXXX<br>XXXXXXX | xxxxx (xxxx, xxxx)<br>xxxxx (xxxx, xxxx) | XX-XXX-XXXX | xx-xxx-xxx | | |

Source Program: xxxxxxx.sas

Table repeats per subject beginning on a new page.

a Adverse events coded with MedDRA Coding Dictionary Version xxx.